CLINICAL TRIAL: NCT05693961
Title: An Invasive Controlled Desaturation Study to Determine the Accuracy of the CART-I Pulse Oximeter (Sky Labs Inc., Korea) in Healthy Adult Volunteers
Brief Title: An Invasive Controlled Desaturation Study to Determine the Accuracy of the CART-I Pulse Oximeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sky Labs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0153
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Healthy
Keywords: Oxygen Saturation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART-I plus (Experimental): CART-I pulse oximeter with a ring-type wearable PPG sensor was placed on each volunteer to evaluate the SpO2 accuracy during steady-state, non-motion conditions.
  Interventions: Device: CART-I plus

INTERVENTIONS:
Device: CART-I plus — CART-I noninvasively measures the oxygen saturation of blood in a local area by screening the bloodstream through the user's finger using PPG signals

SUMMARY:
A pulse oximeter is used for continuous monitoring of peripheral oxygen saturation (SpO2) and plays an important role in the early detection of hypoxia, guiding the titration of supplemental oxygen, and reducing the need for blood gas analysis. Therefore, the SpO2 accuracy of a pulse oximeter should be validated for patient safety. The objective of this study is to evaluate whether the CART-I pulse oximeter with a ring-type wearable PPG sensor (Sky Labs Inc., Seoul, Korea) provides clinically reliable SpO2 readings over the range of 70-100% SaO2, during steady-state, non-motion conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 20-50 years2
* COHb < 3 %
* MetHb < 2 %
* ctHb > 10 g/dl
* Non-smoker
* An individual deemed fit by the investigators to be included in the clinical trial

Exclusion Criteria:

* History of respiratory disease
* History of cardiovascular disease
* Smoker
* Pregnant
* History of fainting
* History of diabetes
* Obesity (defined as BMI > 30 kg/m2)
* Allen's test positive (poor collateral blood supply of hand)
* An individual who is judged to be difficult for the collection of normal PPG signals because CART-I is loose when being worn on fingers other than the thumb and little finger

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-12 (Actual); Primary Completion 2021-06-19 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Accuracy of SpO2 | 1 day
  Mean bias, standard deviation, standard error, maximum/minimum bias, precision are calcuated

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Moon Choi, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Sky Labs, Gyeonggi-do, Pangyo, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luks AM, Swenson ER. Pulse Oximetry for Monitoring Patients with COVID-19 at Home. Potential Pitfalls and Practical Guidance. Ann Am Thorac Soc. 2020 Sep;17(9):1040-1046. doi: 10.1513/AnnalsATS.202005-418FR. PMID 32521167
- [Background] Agarwala P, Salzman SH. Six-Minute Walk Test: Clinical Role, Technique, Coding, and Reimbursement. Chest. 2020 Mar;157(3):603-611. doi: 10.1016/j.chest.2019.10.014. Epub 2019 Nov 2. PMID 31689414
- [Background] Andres-Blanco AM, Alvarez D, Crespo A, Arroyo CA, Cerezo-Hernandez A, Gutierrez-Tobal GC, Hornero R, Del Campo F. Assessment of automated analysis of portable oximetry as a screening test for moderate-to-severe sleep apnea in patients with chronic obstructive pulmonary disease. PLoS One. 2017 Nov 27;12(11):e0188094. doi: 10.1371/journal.pone.0188094. eCollection 2017. PMID 29176802
- [Background] Shiao SY, Ou CN. Validation of oxygen saturation monitoring in neonates. Am J Crit Care. 2007 Mar;16(2):168-78. PMID 17322018